CLINICAL TRIAL: NCT03898765
Title: Dry Blood Spot Screening Test for Biliary Atresia and Other Cholestasis Diseases
Brief Title: Dry Blood Spot Screening Test for Biliary Atresia（DBS-SCReBA）
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XH-BA-1
Record Dates: First submitted 2019-04-01; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Hepatobiliary Disease; Biliary Atresia; Neonatal Cholestasis
Keywords: Dry blood spot test; Biliary Atresia
MeSH Terms: conditions — Digestive System Diseases; Biliary Atresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental：Dry blood spot screening (Experimental)
  Interventions: Diagnostic Test: Dry blood spot screening

INTERVENTIONS:
Diagnostic Test: Dry blood spot screening — Dry blood spot measurement of biomarker for screening biliary atresia

SUMMARY:
Our study aims to develop a screening test for biliary atresia (BA) using dry blood spot to improve patient survival by early diagnosis. Newborn screening dry blood spot will be examined for the direct bilirubin (DB), γ-GT or matrix metalloproteinase-7 (MMP-7) levels. These findings will promote early diagnosis for BA and hence improve the survival.

DETAILED DESCRIPTION:
BA accounts for approximately 60% of the liver transplantations in infants younger than 1 year of age. The diagnosis of BA remains a clinical challenge because affected neonates have signs, symptoms, and serum liver biochemistry that are also seen in those with other causes of neonatal cholestasis.

The success of the Kasai procedure is varied, but a good outcome is correlated with an early diagnosis. Unfortunately, most BA are usually identified later and the average age at surgery is about 60 days. To address this problem, some research groups screen infants for the pale stools or measure bilirubin level in the serum. However, these screening programs have not yet to be implemented because of several reasons. Recently, the relative abundance of serum MMP-7 was suggested to have discriminatory features for infants with BA. Nevertheless, whether the level of MMP-7 elevates in newborn dry blood spot of BA is still undefined. In this study, we will explore a screening strategy based on DB, γ-GT or MMP-7 measurement in newborn screening blood spot, and identify whether DB , γ-GT or MMP-7 measurement in the newborn period could be sensitive and specific for BA.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born in Shanghai

Exclusion Criteria:

* Subjects who do not agree with study protocol
* Subjects who join other clinical trials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Suspected BA | Three to Seven days after birth
  MMP-7 with or without other one or two biomarkers (DB and γ-GT) > upper limit of normal value

CONTACTS AND LOCATIONS:
Overall Officials: Wei Cai, Pro, Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Xinhua Hospital, affiliated to Shanghai Jiao Tong University, School of Medicine, Shanghai, China